CLINICAL TRIAL: NCT00990340
Title: Study to Compare Injection Anxiety Immediately Before the Administration of Each Dose of Tev-Tropin® Between a Needle-syringe Injection Method and a Needle-free Injection Method in Pediatric Subjects With Human Growth Hormone Deficiency
Brief Title: Comparison of a Needle-free Injection Method With a Needle-syringe Injection Method
Acronym: T-jet®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Iris Culbert; Clinical Trials Manager, Teva Neuroscience
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PM201
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-06

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tev-Tropin® needle-free (Active Comparator): needle-free injection method (T-jet®)for 14 days before cross-over to other arm
  Interventions: Device: T-jet® containing TevTropin®
- Tev-Tropin® by Needle-syringe (Active Comparator): needle-syringe injection method for 14 days before cross-over to other arm
  Interventions: Procedure: TevTropin® needle-syringe injection method

INTERVENTIONS:
Device: T-jet® containing TevTropin® — Needle-free delivery method for 14 days before cross-over to other arm
  Other Names: T-jet®
  Arms: Tev-Tropin® needle-free
Procedure: TevTropin® needle-syringe injection method — comparison of delivery methods for 14 days before cross-over to other arm
  Arms: Tev-Tropin® by Needle-syringe

SUMMARY:
The purpose of this study is to obtain psychological response and user preference information on the use of the T jet® device versus the traditional subcutaneous injection administration of Tev Tropin®.

This study will compare subject-reported injection anxiety immediately before the administration of each dose of Tev-Tropin® between a needle-syringe injection method and a needle-free injection method (T-jet®)

DETAILED DESCRIPTION:
The primary efficacy endpoint was the difference in mean subject-reported injection anxiety between the two injection methods as recorded on a 5-point FIS immediately before administration. A higher score denoted greater anxiety.

The injection anxiety score was to be reported by the subject from a row of five faces with values ranging from 5 (the face with the most negative affect) to 1 (the face with the most positive affect).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must require a routine Tev-Tropin® dose that does not exceed 2.5 mg in one injection (0.5 mL) using the dosing schedule individualized for each patient by their prescribing physician
* Male, age 7-17 years, with the capability to provide assent, as determined by the investigator and/or parent or legal guardian
* Clinically definite growth hormone deficiency as previously diagnosed by the investigator or other physician
* Subjects must be using Tev-Tropin® prior to enrollment for 28 days
* Informed consent signed by parent(s) or legal custodian of patient prior to study entry and patient assent as determined by the investigator and/or subject's parent or legal custodian

Exclusion Criteria:

* More than one subcutaneous injection per Tev-Tropin® dose
* Female gender
* Use of any other needle-free injection device at any time
* Current use of another human growth hormone product other than Tev-Tropin®
* Concurrent treatment with other routine injectable medications
* History of benign intracranial hypertension
* Significant communication difficulties, or medical or psychiatric condition, that affects the subject's and/or caregiver's ability to perform the necessary functions to complete the study, or any condition which the investigator in their medical judgment thinks may interfere with participation in the study
* Use of an investigational drug within 30 days prior to randomization
* Contraindications related to routine use of Tev-Tropin® as per investigators' medical judgment (e.g., subjects with closed epiphyses, active proliferative or severe non-proliferative diabetic retinopathy, active malignancy, acute critical illness, or Prader-Willi syndrome who are severely obese or have severe respiratory impairment)
* Current participation in another pharmaceutical or device study
* Previous participation in this study

Ages: 7 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Smith, MD, Study Director — Teva Pharmaceutical Industries, Ltd.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled on 23 September 2009; last subject completed the study on 07 April 2010.
Groups:
- TevTropin® Needle-free Followed by TevTropin® Syringe: needle-free injection method (T-jet®)for 14 days before cross-over to other arm
- TevTropin® by Needle-syringe Followed byTevTropin® Needle-free: needle-syringe injection method for 14 days before cross-over to other arm
Period: First 14-day Treatment
Arm/Group | TevTropin® Needle-free Followed by TevTropin® Syringe | TevTropin® by Needle-syringe Followed byTevTropin® Needle-free
Started | 27 | 25
Completed | 21 | 21
Not Completed | 6 | 4
Not completed — Not Compliant | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 2 | 2
Period: Second 14-day Treatment
Arm/Group | TevTropin® Needle-free Followed by TevTropin® Syringe | TevTropin® by Needle-syringe Followed byTevTropin® Needle-free
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TevTropin® Needle-free Followed by TevTropin® Syringe | TevTropin® by Needle-syringe Followed byTevTropin® Needle-free | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 25 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12.3 (2.31) | 12.5 (2.14) | 12.4 (2.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 25 | 52
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Subject-reported Injection Anxiety Immediately Before Administration
Description: The difference in mean subject-reported injection anxiety between the two injection methods as recorded on a 5 point scale immediately before administration, which scale consisted of a row of five faces with values from 1(most positive)to 5(most negative or greater anxiety.) The score is an average of the Period 1 (Days 1-14) and Period 2 (Days 15-28) assessments; like groups were combined and then averaged. There were 3 visits: Visit 1 (Begin Period 1) Screening and Randomized assignment, Visit 2 (first day of Period 2) Cross over to other assignment, Visit 3 End of Study.
Time Frame: 28 days; Period 1: 14 days, Period 2: 14 days
Population: Of the 52 subjects enrolled, 10 were unevaluable as follows: 4 discontinuations (2 adverse events, 1 lost to follow up, 1 inconsistent participation) 3 non-compliant dosing or diary use, 3 protocol violations ( 2 received devices out of randomized sequence, 1 interruption of injection due to device malfunction.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- TevTropin® Needle-free: Needle-free injection method (T-jet®)for 14 days before cross-over to other arm for 14 days
- TevTropin® by Needle-syringe: Needle-syringe injection method for 14 days before cross-over to other arm for 14 days
Arm/Group | TevTropin® Needle-free | TevTropin® by Needle-syringe
Number analyzed (Participants) | 42 | 42
Scores on a scale | 2.15 (1.019) [44.6 to 60.7] | 1.98 (1.024) [38.7 to 54.9]

2. Secondary Outcome: Subject-reported Injection Pain Immediately Following Administration.
Description: as for outcome 1
Time Frame: 28 days; Period 1: 14 days, Period 2: 14 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | TevTropin® Needle-free | TevTropin® by Needle-syringe
Number analyzed (Participants) | 42 | 42
Scores on a scale | 0.96 (0.994) | 0.89 (1.015)

3. Secondary Outcome: Subject or Caregiver Reported Perception of Ease of Preparation as Recorded Weekly on a 5-point Scale.
Description: The difference in mean subject-reported injection anxiety between the two injection methods as recorded on a 5 point scale immediately before administration, which scale consisted of a row of five faces with values from 1(most positive)to 5(most negative or greater anxiety.) The score is an average of the Period 1 (Days 1-14) and Period 2 (Days 15-28) assessments; like arms were combined and then averaged. There were 3 visits: Visit 1 (Begin Period 1) Screening and Randomized assignment, Visit 2 (first day of Period 2) Cross over to other assignment, Visit 3 End of Study.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | TevTropin® Needle-free | TevTropin® by Needle-syringe
Number analyzed (Participants) | 42 | 42
Scores on a scale | 2.55 (1.222) | 1.78 (0.967)

4. Secondary Outcome: Subject or Caregiver Reported Perception of Ease of Administration as Recorded Weekly on a 5-point Scale.
Description: The difference in subject-reported overall satisfaction between the two injection methods as recorded on a 5-point scale following the end of each period of the study. The overall satisfaction was to be rated by the subject on a 5-point scale as 1 (Really Unhappy) to 5 (Really Happy), a higher score denoting greater satisfaction. Overall satisfaction is obtained only once at the end of each period; Period 1 Tjet group was added to Period 2 Tjet group and Period 1 syringe group was added to Period 2 syringe group; no averaging was necessary.
Time Frame: 28 Days; end of Period 1(14 days) and end of Period 2 (14 days)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | TevTropin® Needle-free Followed by TevTropin® Syringe | TevTropin® by Needle-syringe Followed byTevTropin® Needle-free
Number analyzed (Participants) | 42 | 42
Scores on a scale | 2.40 (1.246) | 1.76 (1.052)

5. Secondary Outcome: Subject-reported Overall Satisfaction Following the End of Each Period of the Study.
Description: as for outcome 4
Time Frame: 28 Days; end of Period 1(14 days) and end of Period 2 (14 days)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | TevTropin® Needle-free | TevTropin® by Needle-syringe
Number analyzed (Participants) | 42 | 42
Scores on a scale | 3.31 (1.339) | 3.96 (1.147)

ADVERSE EVENTS:
Arm/Group | TevTropin® Needle-free Followed by TevTropin® Syringe | TevTropin® by Needle-syringe Followed byTevTropin® Needle-free
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.